CLINICAL TRIAL: NCT07112378
Title: A Randomized Study Evaluating 2 Dose Regimens of Dupilumab in Children ≥6 Months of Age Weighing ≥5 to <15 kg With Active Eosinophilic Esophagitis
Brief Title: A Study of Dupilumab in Small Children With an Allergic Condition of the Esophagus (Food Pipe): Eosinophilic Esophagitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R668-EE-2423
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: Type 2 Inflammatory; Allergic/immune-mediated; Esophageal dysfunction
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Diseases | interventions — dupilumab

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosing Regimen 1 (Experimental)
  Interventions: Drug: dupilumab
- Dosing Regimen 2 (Experimental)
  Interventions: Drug: dupilumab

INTERVENTIONS:
Drug: dupilumab — Administered as defined in the protocol
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
This study is researching an experimental drug called dupilumab (called "study drug"). The study is focused on children with active eosinophilic esophagitis (EoE; an inflammatory disease of the esophagus) which impacts feeding and nourishment.

The aim of the study is to see how safe, tolerable, and effective the study drug is when given for 24 weeks to children with active EoE.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Pediatric patients aged ≥6 months and weighing ≥5 kg and <15 kg at screening with active EoE
2. History of symptom(s) determined by the investigator to be the result of EoE in the month prior to screening, as defined in the protocol
3. Baseline endoscopic biopsies, performed during the screening period, with a demonstration on central reading of intraepithelial eosinophilic infiltration in at least 2 of the 3 biopsied esophageal regions, as defined in the protocol

Key Exclusion Criteria:

1. Prior participation in a dupilumab clinical trial or past or current treatment with dupilumab
2. Initiation or change of a food-elimination diet regimen or re-introduction of a previously eliminated food group in the 6 weeks prior to screening. Patients on a food-elimination diet must remain on the same diet throughout the study
3. Other causes of esophageal eosinophilia or the following conditions: eosinophilic gastroenteritis, hypereosinophilic syndrome, and eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome)
4. Active Helicobacter pylori infection
5. History of Crohn's disease, ulcerative colitis, celiac disease, or prior esophageal surgery
6. Any esophageal stricture unable to be passed with a standard, diagnostic, upper endoscope or any critical esophageal stricture that requires dilation at screening
7. History of bleeding disorders or esophageal varices that, in the opinion of the investigator, would put the patient at undue risk for significant complications from an endoscopic procedure
8. Treatment with swallowed topical corticosteroids within 8 weeks prior to baseline standard of care endoscopy

NOTE: Other Protocol-Defined Inclusion/Exclusion Criteria Apply

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-08-21 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Serious Adverse Events (SAEs) | Up to 24 Weeks

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) leading to permanent discontinuation of study treatment | Up to 24 Weeks
Incidence of treatment-emergent Adverse Event of Special Interest (AESIs) | Up to 24 Weeks
Incidence of TEAEs | Up to 24 Weeks
Proportion of patients achieving peak esophageal intraepithelial eosinophil count of ≤6 eosinophils per high power field (eos/hpf) (400×) | At Week 24
Proportion of patients achieving peak esophageal intraepithelial eosinophil count of <15 eos/hpf (400×) | At Week 24
Percent change in peak esophageal intraepithelial eosinophil count (eos/hpf) | Baseline to Week 24
Change in body weight for age percentile | Baseline up to Week 24
Concentrations of functional dupilumab in serum | Baseline up to Week 24
Incidence of Anti-Drug Antibody (ADA) to dupilumab | Up to Week 36
Titer of ADA to dupilumab | Up to Week 36
Incidence of Neutralizing Antibody (NAb) to dupilumab | Up to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (5):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - GI Care for Kids LLC, Atlanta, Georgia
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina, Bioinformatics Building, Chapel Hill, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/